CLINICAL TRIAL: NCT04796519
Title: A Comparison of Balance and Fall Risk in Patients With Unilateral and Bilateral Total Knee Arthroplasty
Brief Title: Comparison of Balance and Fall Risk in Unilateral and Bilateral Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Erman tütüncüler, Research assistant, Pamukkale University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Balance, Fall risk after TKA
Record Dates: First submitted 2021-03-04; First posted 2021-03-15 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Knee Arthropathy
Keywords: fall risk; balance; total knee arthroplasty; function
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unilateral TKA (Experimental): Unilateral total knee arthroplasty group (UTKA) consisted of patients who did not undergo a second TKA within 3 months of the first TKA
  Interventions: Procedure: Total knee arthroplasty
- Bilateral TKA (Experimental): bilateral total knee arthroplasty group (BTKA) were those who had a second TKA within 12 months after initial TKA
  Interventions: Procedure: Total knee arthroplasty

INTERVENTIONS:
Procedure: Total knee arthroplasty — Surgical procedure

SUMMARY:
Static or dynamic postural control cannot be fully restored in patients with Total Knee Arthroplasty (TKA). Moreover, deficits in balance and postural control may still be present in both extremity after TKA. However, the contralateral knee OA grade, asymmetrical gait pattern, and postural sways still remain a risk factor for balance deficits and falls. Based on this rationale, the aim of this study is to evaluate the balance and fall risk before and after TKA in patients who suffered from bilateral knee osteoarthritis and to clarify the balance and fall risk difference between unilateral and bilateral TKA patients.

DETAILED DESCRIPTION:
Falls are one of the leading causes of increased morbidity and mortality in the elderly population and are substantial contributor to increase healthcare cost burden. Pain, strength deficits, knee joint deformities, balance and proprioceptive impairments associated with severe knee OA, contribute to an increased risk of falling among elderly, and more than 50% of this population experience a fall each year. Static or dynamic postural control cannot be fully restored in patients with Total Knee Arthroplasty (TKA). Moreover, deficits in balance and postural control may still be present in both extremity after TKA. Increased weight-bearing on the operative side after TKA and reduced weight-bearing weight in the contralateral osteoarthritic knee can reduce pain and improve balance-related functions. However, the contralateral knee OA grade, asymmetrical gait pattern, and postural sways still remain a risk factor for balance deficits and falls. Based on this rationale, the aim of this study is to evaluate the balance and fall risk before and after TKA in patients who suffered from bilateral knee osteoarthritis and to clarify the balance and fall risk difference between unilateral and bilateral TKA patients.

ELIGIBILITY:
Inclusion Criteria:

* age between 55 to 85 years, patients with bilateral osteoarthritis, Kellgren-Lawrence grade 3-4, patients capable of understanding verbal and written instructions.

Exclusion Criteria:

* revision TKA surgery, American Society of Anesthesiologists score >3, neurologic compromise, psychiatric problems, regular hypnotic and/or anxiolytic medication usage, dementia.

Ages: 46 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-10-10 (Actual)

PRIMARY OUTCOMES:
Fall risk evaluation | 3 months
  Fall risk was evaluated using the Biodex Balance System SD (Biodex Medical Systems Inc., Shirley, NY, USA). The Fall Risk test was conducted to identify potential fall candidates. Test results are compared with age-related normative data.
Balance evaluation | 3 months
  Balance (Postural Stability and Sensory Integration) was evaluated using the Biodex Balance System SD (Biodex Medical Systems Inc., Shirley, NY, USA). Postural Stability Test was applied to determine a patient's ability to maintain the centre of balance. Sensory Integration Test aims to evaluate the individual's ability to both integrate various senses to maintain balance and to compensate when one of these senses is missing. This test included four conditions: Eyes Open-Firm Surface, Eyes Closed-Firm Surface, Eyes Open-Foam Surface, and Eyes Closed-Foam Surface. Each assessment lasted 30 seconds, with 10 seconds of rest in between assessments.

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index score | 3 months
  It is a patient reported questionnaire that evaluates pain, stiffness, and physical function in patients with hip and knee OA. The index consists of 24 questions and is completed in less than 5 minutes. The scores of the questions range from 0 (none) to 4 (very severe) and the results are evaluated over 100 points (minimum score:0 and the maximum score:100). Higher scores indicates worst knee functions.
Quality of life measure | 3 months
  Patients' quality of life were evaluated with Short Form-12 for seconder outcome. Higher scores indicates better quality of life.
Sit-to-stand test | 3 months
  The patient was seated in the middle of a chair with a height of 44 cm, with his back straight, arms crossed in front of his chest, and feet on the ground. The patient was asked to get up from the chair and sit down as much as the patient could for 30 seconds. The exact number of starts made formed the patient's score. Higher scores indicates better overall strength.
9-step stair climbing test | 3 months
  The patient was asked to climb and descend the 9-step 16-20 centimeter ladder as quickly but safely as possible. The patient was allowed to use a handrail or a walking aid, and the method used was recorded. The test was started with the start command and the time stopped when the patient returned to the starting place. The patient was allowed to stop and rest when requested, but the duration was continued. The total time was recorded as a score. Lower scores indicates better knee functions.
40 m fast-paced walk test | 3 months
  Patients were asked to walk along the 10-meter track without running but as fast as possible, turn around the cone at the finish, and complete the 40-meter total distance. After the patient passed the baseline in the last stage, the time was stopped and the total time was recorded. Lower scores indicates better walking capacity.

CONTACTS AND LOCATIONS:
Overall Officials: Erman Tütüncüler, Dr., Principal Investigator — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zora H, Gungor HR, Bayrak G, Savkin R, Buker N. Does mini-midvastus approach have an advantageous effect on rapid recovery protocols over medial parapatellar approach in total knee arthroplasty? Jt Dis Relat Surg. 2020;31(3):571-581. doi: 10.5606/ehc.2020.76387. PMID 32962591
- [Result] Vala CH, Karrholm J, Kanis JA, Johansson H, Sten S, Sundh V, Karlsson M, Lorentzon M, Mellstrom D. Risk for hip fracture before and after total knee replacement in Sweden. Osteoporos Int. 2020 May;31(5):887-895. doi: 10.1007/s00198-019-05241-x. Epub 2019 Dec 12. PMID 31832694
- [Result] Bakirhan S, Angin S, Karatosun V, Unver B, Gunal I. Physical performance parameters during standing up in patients with unilateral and bilateral total knee arthroplasty. Acta Orthop Traumatol Turc. 2012;46(5):367-72. doi: 10.3944/aott.2012.2684. PMID 23268822